CLINICAL TRIAL: NCT02373579
Title: Effect of Omega-3 Fatty Acids on Methotrexate Induced Hepatotoxicity in Children With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nancy Samir Elbarbary (Other)
Responsible Party: Sponsor-Investigator, Nancy Samir Elbarbary, Assistant professor, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ain Shams University 1351
Record Dates: First submitted 2015-02-02; First posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: omega-3 fatty acids; methotrexate; hepatotoxicity
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Fatty Acids, Omega-3; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention arm with Omega 3 FA (Active Comparator): included standard risk ALL pediatric patients who were supplemented with oral omega-3 capsule (one capsule / day) .
  Omega-3 was supplied as soft gelatin capsules in a dose of 1000 mg of omega-3 fatty acids/day .
  Interventions: Drug: Omega-3 Fatty Acids; Drug: Methotrexate
- control group (Active Comparator): control group, included pediatric patients with standard risk acute lymphoblastic leukemia in maintenance phase day 0 and receiving oral Methotrexate (20 mg / m2) weekly without any supplementation .
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Omega-3 Fatty Acids — study group, included standard risk ALL pediatric patients who were supplemented with oral omega-3 capsule (one capsule / day) .
  Omega-3 was supplied as soft gelatin capsules in a dose of 1000 mg of omega-3 fatty acids/day .
  Other Names: Super-omega®
  Arms: Intervention arm with Omega 3 FA
Drug: Methotrexate — control group, included pediatric patients with standard risk acute lymphoblastic leukemia in maintenance phase day 0 and receiving oral Methotrexate (20 mg / m2) weekly without any supplementation .
  Other Names: Rheumatrex

SUMMARY:
Study the role of oxidative stress in methotrexate induced hepatic damage, and the possible protective effect of OMEGA-3 fatty acids against methotrexate hepatotoxicity using clinical and biochemical parameters.

DETAILED DESCRIPTION:
The patients were divided into two groups :Group I: control group, included pediatric patients with standard risk acute lymphoblastic leukemia in maintenance phase day 0 and receiving oral Methotrexate (20 mg / m2) weekly without any supplementation .

Group II: study group, included standard risk ALL pediatric patients who were supplemented with oral omega-3 capsule (one capsule / day) .

Omega-3 was supplied as soft gelatin capsules in a dose of 1000 mg of omega-3 fatty acids/day . This is in addition to chemotherapy from day one of maintenance phase receiving oral Methotrexate (20 mg / m2) Weight -adjusted doses on days 8, 15, 22, 29,36,43,50,57,64,71and 78).

Both groups were followed up for six months . All patients were under free diet and were maintained on standard diet throughout the study ( 6 months). None of them were on regular vitamin supplementation before diagnosis or at time of chemotherapy administration.

Patients follow up:

The patients were followed up every three week for the whole study period for assessing the effect and compliance to both MTX and Omega-3 fatty acid and for monitoring any potential adverse effect.

Group I were asked on each visit about signs of hepatic toxicity ( fatigue , weakness , loss of appetite , vague abdominal pain , color of urine and sclera and jaundice ), their laboratory results were revised to know level of ALT as a marker of liver injury .

Group II were asked on each visit about signs of hepatotoxicity , their laboratory data were revised , any side effects resulted from use Omega-3 fatty acids:

(increased bleeding tendency, fishy smell , nausea , diarrhea , or if there is any relapses occurred , and to be sure that the patients were compliant to prescribed medication.

Investigations:

Blood samples were collected from every patient at day 0 of maintenance and after six months for estimation of Malondialdehyde (MDA), Total antioxidant capacity (TAC), super oxide dismutase ,liver function tests and uric acids . Blood was collected into heparinised tubes which were protected from light and processed immediately after sampling. At the time of collecting the blood samples, patients were free of any potentially confounding or interfering conditions, such as infections or fever.

ELIGIBILITY:
Inclusion Criteria:

* Child age: less than 17 years old.
* Taking oral methotrexate in maintenance therapy.
* Patients are at cycle one day zero.

Exclusion Criteria:

* Child infected by hepatitis B or C viruses.
* Child taking medications or having a condition causing elevation in liver enzymes level other than methotrexate.(eg:thrombosis ,antibiotic therapy, infiltrating malignancy ,auto immune manifestations or having TPN)
* Child remission.
* Child death
* Child drop out due to non compliance

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2012-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability by measuring Malondialdehyde (MDA) level changes . | six months
Number of Participants with Adverse Events as a Measure of Safety and Tolerability by measuring Total antioxidant capacity (TAC) level changes. | six months
Number of Participants with Adverse Events as a Measure of Safety and Tolerability by measuring superoxide dismutase (SOD) level changes. | six months
Number of Participants with Adverse Events as a Measure of Safety and Tolerability by measuring uric acids levels changes . | Six months

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability by measuring ALT value changes. | six months

REFERENCES:
- [Derived] Elbarbary NS, Ismail EA, Farahat RK, El-Hamamsy M. omega-3 fatty acids as an adjuvant therapy ameliorates methotrexate-induced hepatotoxicity in children and adolescents with acute lymphoblastic leukemia: A randomized placebo-controlled study. Nutrition. 2016 Jan;32(1):41-7. doi: 10.1016/j.nut.2015.06.010. Epub 2015 Jul 17. PMID 26421385